CLINICAL TRIAL: NCT04273893
Title: A Pilot Randomized Study of Lymphocyte Depletion & Change in Lymphocyte Functionality During Lung Stereotactic Body Radiation (SBRT) Therapy Treatment by Selectively Reducing Irradiation of Immune Rich Organs Compared to Standard of Care Control Group
Brief Title: Lymphocyte Depletion and Change in Lymphocyte Functionality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Krishni Wijesooriya, Professor of Radiation Oncology - Medical Physics, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21718; 5R01CA234281-03 (NIH)
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lymphocyte Depletion
Keywords: Lymphocyte Depletion and Change; SBRT; NSCLC; Lung Cancer; radiation therapy; non small cell; Stereotactic body radiation therapy; Treatment related lymphopenia
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants, clinical research staff, and treating clinicians will be aware of arm assignment. The labels on research blood will not include the treatment arm on which the participant is assigned and this information will not be provided to lab investigators and staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT Additional treatment planning dose optimization (Experimental): Lung SBRT 50-60Gy in 5 fractions with standard of care planning and additional treatment planning dose optimization criteria to minimize decrease in lymphocyte count beyond dosimetric criteria from RTOG 0915/0813 SBRT trials.
  Interventions: Radiation: SBRT with additional treatment planning dose optimization; Diagnostic Test: Blood Draws
- SBRT with standard of care planning only (Active Comparator): Lung SBRT 50-60Gy in 5 fractions with standard of care planning (no additional dose optimization beyond SOC)
  Interventions: Radiation: SBRT with standard of care planning only; Diagnostic Test: Blood Draws

INTERVENTIONS:
Radiation: SBRT with additional treatment planning dose optimization — Lung SBRT 50-60Gy in 5 fractions with standard of care planning and additional treatment planning dose optimization criteria to minimize decrease in lymphocyte count beyond dosimetric criteria from RTOG 0915/0813 SBRT trials.
  Arms: SBRT Additional treatment planning dose optimization
Radiation: SBRT with standard of care planning only — Lung SBRT 50-60Gy in 5 fractions with standard of care planning (no additional dose optimization beyond SOC)
  Arms: SBRT with standard of care planning only
Diagnostic Test: Blood Draws — CBC w/ Diff and additional blood analysis for all participants in both groups. Blood draws will prior to treatment, end of treatment, 4 weeks after treatment, and 6 months after treatment.

SUMMARY:
Lymphocytes are a type of white blood cell (WBC) responsible for adaptive immunity. Thoracic tumors are adjacent to many blood/immune rich organs including the great vessels, heart, thoracic-spine, and lymph-node-stations. During radiation treatment the impact to lymphocytes can be significant. This may cause a decrease in the amount of lymphocytes. A researcher at UVA has created a system to predict and reduce the immune cell reduction following lung SBRT treatments beyond standard of care. The predicted decrease in lymphocytes will be compared to the actual decrease in lymphocytes found in peripheral blood.

Researchers have found a way to give radiation that they think will result in a smaller decrease in lymphocytes after radiation. There will be two groups in this study, about half of the participants will have their radiation designed to decrease radiation to organs with a lot of blood and the other half will receive standard radiation therapy.

Participants are being asked to take part in this study because the participants have been diagnosed with NSCLC and will be receiving a type of radiation therapy called stereotactic body radiation therapy (SBRT) where high doses of radiation will be delivered to the tumor, while minimizing damage to healthy surrounding tissues.

DETAILED DESCRIPTION:
Lymphocytes play a crucial role in the body's response to cancer by directly attacking tumors, inhibiting tumor growth and spread, and detecting and potentially eliminating emerging tumors. Tumor-infiltrating lymphocytes (TILs) are commonly found within tumors, and studies have shown that their presence is associated with more favorable outcomes. Radiation therapy (RT), particularly Stereotactic Body Radiation Therapy (SBRT), modulates the immune system by promoting the generation of Cytotoxic T Lymphocytes (CTLs) and enhancing T cell infiltration into tumors. These CTLs may eliminate distant metastases or residual disease (abscopal effect) not targeted by the primary treatment.

Lymphopenia, a known consequence of radiation therapy to virtually every part of the body, was first described in the early 20th century shortly after the discovery of X-rays. It is highly possible that irradiation of blood rich and lymphatic rich organs and bone marrow would reduce the lymphocyte counts significantly.

Additionally, recent data have suggested that lymphocyte subsets exhibit differential sensitivity to radiation, with helper CD4+ T cells being more sensitive than cytotoxic CD8+ T cells in glioblastoma (GBM) treated with RT and temozolomide, and naïve T cells more sensitive than memory T cells in prostate cancer.

Based on existing data on the effects of irradiation on total lymphocyte count and the effects on subsets of T cells, the investigators have created a lymphodepletion predictive algorithm. In this clinical trial, the investigators will test whether optimized SBRT plans lead to lower lymphocyte depletion and whether the algorithm can accurately predict lymphocyte decreases following SBRT. Optimized SBRT plans will meet all standard of care dose-volume objectives for SBRT and for the protection of organs-at-risk (OAR), but will also minimize radiation exposure to circulating blood and lymphatics, including the heart, great-vessels, lymph-node-stations, and thoracic-spine beyond what is currently optimized to reduce the integral dose to circulating blood/lymphocytes. This study will allow us to evaluate the performance of our predictive algorithm for post-SBRT decrease in lymphocyte count and to determine whether additional steps in SBRT planning will deliver lower risk of post-SBRT decreases in lymphocyte count.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide written informed consent and to comply with the study protocol.
2. Diagnosis of biopsy confirmed non-small cell lung cancer (NSCLC) with planned treatment with SBRT as definitive therapy OR imaging confirmed lung lesion for which SBRT is planned for primary lung cancer (when clinician determines biopsy is not indicated), Registration should occur within 5 business days (before or after) of planning CT.
3. Patients must decline surgery or tumor(s) must be considered to be medically inoperable
4. Location and size of tumor- Participants must have either:

   * peripherally located tumors (> 2 cm in all directions from the proximal bronchial tree; see Figure 2 above) as defined by RTOG 0915, OR
   * centrally located tumors (tumor size ≤ 5 cm, tumors within or touching the zone of the proximal bronchial tree or adjacent to mediastinal or pericardial pleura) as defined by RTOG 0813.
5. Patients with recurrence of prior surgically treated lung cancers are eligible if no further surgery is planned and they otherwise meet the eligibility criteria.
6. Measurable disease on chest CT, PET CT, CT simulation at diagnosis ( must be within 8 weeks of SBRT).
7. Pre- radiation therapy total lymphocyte count > 0.5k/μL on blood count drawn within 2 weeks prior to registration.
8. In the opinion of the treating clinician, patient is medically able to tolerate the study SBRT treatment of 50-60 Gy in 5 fractions.
9. ECOG performance status of 0-2.
10. Age ≥ 18 years.
11. If participant is a woman of childbearing potential (WOCBP), agreement to adhere to contraception requirements from the time of consent through completion of SBRT.

Exclusion Criteria

1. Prior history of radiation therapy within 2 years of registration, however radiation therapy for skin cancer is allowed
2. Systemic anti-cancer therapy within the last year prior to registration or planned use during or within 6 months following SBRT.
3. Major surgery within the last 30 days before registration and/or planned before the completion of the 6 months post SBRT follow up timeframe.
4. Subject is a prisoner.
5. Subject is a pregnant woman.
6. Patient is not medically able to tolerate the study SBRT treatment of 50-60 Gy in 5 fractions or cannot comply with other aspects of the study including serial bloodwork.
7. Subject has HIV, AIDS, any type of hepatitis and/or any blood borne infectious disease for which the research lab cannot receive blood samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2025-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Krishni Wijesooriya, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijesooriya K, Nguyen C, Conaway MR, Read PW, Romano K, Lum LG, Thakur A, Lain DW, McLaughlin CM, Luminais CK, Wood S, Williams G, Chen J, Walker B, Sprouts D, Muller D, Ward K, Dutta S, Sanders J, Cousins D, Asare E, Nesbit E, Chavis YC, Walker KV, Janowski E, Showalter T, Larner JM. First Measurement: Proactive Immune Cell Sparing in Radiation Therapy. medRxiv [Preprint]. 2025 Jan 6:2025.01.05.25320011. doi: 10.1101/2025.01.05.25320011. PMID 39830271

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at one academic medical center between February 2020 and April 2023. Participants were randomized with equal allocation to each ordering (optimize SBRT ARM or Standard SBRT ARM) using a stratified block randomization scheme with varying block sizes. Randomization occurred prior to start of treatment.
Pre-assignment Details: Two participants were discontinued from the study before treatment but after randomization. One participant became ineligible after discovering new medical history information and the other participant withdrew consent.
Period: Overall Study
Arm/Group | SBRT Additional Treatment Planning Dose Optimization | SBRT With Standard of Care Planning Only
Started | 26 | 27
Completed Treatment | 25 | 26
Completed 4 Week Follow Up | 25 | 25
Completed | 24 | 19
Not Completed | 2 | 8
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Treatment of Disease Progression | 0 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two participants were discontinued from the study before staring treatment but after randomization. One participant became ineligible after discovering new medical history information and the other participant withdrew consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT Additional Treatment Planning Dose Optimization | SBRT With Standard of Care Planning Only | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 22 | 23 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 24 | 27 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55
Lung Lesion Location [Count of Participants; unit: Participants]
  Central | 9 | 6 | 15
  Peripheral | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Impact of Lymphocyte-Sparing SBRT Planning Objectives on Post-SBRT Lymphocyte Count
Description: Mean percentage difference of measured absolute lymphocyte counts between the baseline and at each time points for the two separate arms
Time Frame: Baseline to End of SBRT (up to 12 days), 4 weeks after SBRT (up to 1.5 months) and 6 months after SBRT (up to 10 months)
Population: Participants completing the CBC with Differential lab test to obtain absolute lymphocyte count results. A few participants missed the lab test or discontinued from the study for various reason resulting no lab data for a particular timepoint.
Measure: Mean (Standard Deviation); unit: Percentage from baseline
Arm/Group | SBRT Additional Treatment Planning Dose Optimization | SBRT With Standard of Care Planning Only
Number analyzed (Participants) | 25 | 26
Percentage from baseline
  Between Baseline and End of SBRT | -15 (18) | -30 (21)
  Between Baseline and 4 weeks after SBRT: number analyzed (Participants) | 25 | 25
  Between Baseline and 4 weeks after SBRT | -22 (24) | -34 (18)
  Between Baseline and 6 months after SBRT: number analyzed (Participants) | 24 | 22
  Between Baseline and 6 months after SBRT | -15 (29) | -24 (22)
Statistical Analysis 1: Comparison: SBRT Additional Treatment Planning Dose Optimization vs SBRT With Standard of Care Planning Only; Test type: Other; p = 0.05, t-test, 2 sided — Changes from baseline ALC were conducted using repeated measures models with an unstructured covariance matrix and model terms for tumor location, follow-up time. Adjustments for stratification factors were made using least squares means

2. Primary Outcome: Determine if an Algorithm Can Predict the Magnitude of Post SBRT Lymphocyte Depletion Prospectively for Participants With NSCLC
Description: Median of the difference between predicted value and observed measurement of lymphocyte absolute counts.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: 10^9 cell/L
Arm/Group | SBRT Additional Treatment Planning Dose Optimization | SBRT With Standard of Care Planning Only
Number analyzed (Participants) | 25 | 26
10^9 cell/L
  End of SBRT | 0.14 [0.06 to 0.27] | 0.18 [0.08 to 0.38]
  4 Weeks after SBRT: number analyzed (Participants) | 25 | 25
  4 Weeks after SBRT | 0.27 [0.18 to 0.40] | 0.18 [0.08 to 0.30]
  6 Months after SBRT: number analyzed (Participants) | 23 | 22
  6 Months after SBRT | 0.23 [0.14 to 0.41] | 0.21 [0.14 to 0.46]

ADVERSE EVENTS:
Time Frame: From the time informed consent is obtained until 6 months after completion of SBRT (up to 11months)
Arm/Group | SBRT Additional Treatment Planning Dose Optimization | SBRT With Standard of Care Planning Only
All-Cause Mortality (participants affected / at risk) | 1/26 | 2/27
Serious Adverse Events (participants affected / at risk) | 10/26 | 7/27
Other Adverse Events (participants affected / at risk) | 24/26 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT Additional Treatment Planning Dose Optimization (N=26) | SBRT With Standard of Care Planning Only (N=27)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 5 (5) | 4 (4)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Electrolyte Imbalance
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) — Bloody Diarrhea
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT Additional Treatment Planning Dose Optimization (N=26) | SBRT With Standard of Care Planning Only (N=27)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) — Chest Tightness
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (10)
Edema limbs (General disorders) | 3 (3) | 4 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1) — Cold intolerance
Fatigue (General disorders) | 8 (8) | 9 (9)
Fever (General disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) — Rib Fracture
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — knee pain and swelling
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — inflammatory changes in lung
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchiolectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT04273893/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04273893/ICF_002.pdf